CLINICAL TRIAL: NCT06989918
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy of MHB018A Injection in Subjects With Active Moderate-to-Severe Thyroid Eye Disease.
Brief Title: MHB018A Treatment in Patients With Active Thyroid Eye Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Minghui Pharmaceutical (Hangzhou) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHB018A-P-301
Record Dates: First submitted 2025-05-09; First posted 2025-05-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Associated Ophthalmopathies
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MHB018A (Experimental): 6 subcutaneous injections of MHB018A, 450mg once every 4 weeks (q4w)
  Interventions: Drug: MHB018A
- MHB018A Placebo (Placebo Comparator): 6 subcutaneous injections of MHB018A placebo once every 4 weeks (q4w)
  Interventions: Drug: MHB018A placebo

INTERVENTIONS:
Drug: MHB018A — MHB018A 450mg for subcutaneous injection once every 4 weeks (Q4W)
  Arms: MHB018A
Drug: MHB018A placebo — 6 subcutaneous injections of MHB018A placebo once every 4 weeks (q4w)
  Arms: MHB018A Placebo

SUMMARY:
The primary objective of this study is to investigate the efficacy, safety, and tolerability of MHB018A, a humanized anti-IGF1R antibody, administered q4W for 6 months, in comparison to placebo, in the treatment of participants suffering from active TED.

DETAILED DESCRIPTION:
The percentage of subjects with a reduction in proptosis of ≥2 mm in the study eye/target eye compared to baseline, without deterioration (≥2 mm) in the fellow eye.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participating in the study and signing the informed consent form;
2. Aged 18-75 years (inclusive), of any gender;
3. Clinical diagnosis of active Thyriod Eye Disease (TED). The Clinical Activity Score (CAS) of the study eye/target eye at screening and baseline must be ≥3 points (7-point scale).
4. Subjects with a clinical diagnosis of moderate to severe TED at screening and baseline.
5. Does not require immediate surgical ophthalmological intervention, and no corrective surgery/orbital radiotherapy is planned during the study.
6. Diabetic subjects must have well-controlled stable disease.
7. Sufficient bone marrow and organ function.
8. Eligible subjects of childbearing potential (male and female) must agree to use reliable contraceptive methods; female subjects of childbearing potential must have a negative blood pregnancy test within 7 days before the first use of the study drug and must not be breastfeeding.
9. Subject is willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the study.

Exclusion Criteria:

1. Decreased best corrected visual acuity due to optic neuropathy as defined by a decrease in vision within the last 6 months of two lines of Snellen chart, new visual field defect or color defect secondary to optic nerve involvement.
2. Corneal decompensation unresponsive to medical management.
3. Decrease in CAS of ≥ 2 points or decrease in proptosis of ≥ 2 mm between screening and baseline.
4. Free thyroxine (FT4) and free triiodothyronine (FT3) levels <50% above or below the normal reference range at screening.
5. Subjects who have previously received orbital radiotherapy or ophthalmic surgery for TED.
6. Subjects who received oral or intravenous corticosteroids or corticosteroid eye drops/ointments for TED within 4 weeks before the first dose; subjects who received periorbital/orbital steroid injections within 3 months before the first dose.
7. Subjects who used oral or intravenous corticosteroids for reasons other than TED within 4 weeks prior to Screening, excluding local use (topical, nasal, inhalation).
8. Any previous treatment with rituximab, tocilizumab, other immunosuppressive agent use within 3 months prior to Screening.
9. Previous treatment targeting IGF-1R.
10. Selenium and biotin must be discontinued 3 weeks prior to Screening and must not be restarted during the trial; however, taking a multivitamin that includes selenium and/or biotin is allowed.
11. Use of an investigational agent for any condition within 30 days prior to Screening or anticipated use during the course of the trial.
12. Identified pre-existing ophthalmic disease that, in the judgment of the Investigator, would preclude study participation or complicate interpretation of study results.
13. Malignant condition in the past 5 years before signing the ICF (except successfully treated basal/squamous cell carcinoma of the skin).
14. Acute cardiovascular disease history or treatment within 6 months before the first dose.
15. Presence of poorly controlled hypertension with systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg; Renal artery stenosis.
16. Pregnant or lactating women.
17. Drug or alcohol abuse during the screening period.
18. Hearing impairment history in either ear during the screening period; or abnormal pure tone audiometry results.
19. Biopsy-proven or clinically suspected inflammatory bowel disease.
20. Positive results for serum virology tests (defined as pos
21. Subjects who received or planned to receive live or attenuated live vaccines within 4 weeks before the first dose or during the study period.
22. Subjects who underwent major surgery within 4 weeks before the first dose or are expected to undergo surgery during the study period or within 4 weeks after the study.
23. Known hypersensitivity to any of the components of MNB018A or prior hypersensitivity reactions to mAbs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Proptosis Responder Rate at Week 24 | Week 24
  The percentage of subjects with a reduction in proptosis of ≥2 mm in the study eye/target eye compared to baseline, without deterioration (≥2 mm) in the fellow eye.

SECONDARY OUTCOMES:
Overall response rate | Week 24
  The percentage of subjects with ≥2-points in Clinical Activity Score (CAS) reduction and ≥2 mm reduction in proptosis from baseline, provided there is no corresponding deterioration (≥2-points/mm increase) in CAS or proptosis in the fellow eye.
Change in proptosis | Baseline, up to Week 24
  Change from baseline in proptosis in the study eye as measured by exophthalmometer at Week 24
Percentage of subjects with CAS of 0 or 1 | Week 24
  The percentage of subjects with a CAS of 0 or 1 in the study eye/target eye.
Change in CAS | Week 24
  The mean change from baseline to Week 24 in the CAS in the study eye/target eye.
Diplopia response rate | Week 24
  The percentage of subjects with a reduction in diplopia severity by ≥1 grade.
Change in Quality of Life (GO-QOL) Scores | Week 24
  The mean change in scores from the Graves' Ophthalmopathy Quality of Life questionnaire compared to baseline.
Pharmacokinetic Parameter Trough Concentration for MHB018A | Up to Week 24
  Trough concentration (Ctrough) will be assessed using non-compartmental methods in participants randomized to the MHB018A group.
Anti-MHB018A antibody (ADA) incidence | Up to Week 24 and at end-of-trial (EOT) visit
  The percentage of subjects developing anti-MHB018A antibodies.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China